CLINICAL TRIAL: NCT05884593
Title: Analysis of Pedicle Screw Accuracy to Plan Using Medtronic Mazor Robotic System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Andrew Grossbach, Assistant Clinical Professor Residency Program Director Deformity and Robotic Spinal Fellowship Director, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020H0434
Record Dates: First submitted 2023-03-15; First posted 2023-06-01 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Spinal Deformity; Spinal Infection; Trauma; Neoplastic Processes; Degenerative Spinal Conditions
MeSH Terms: conditions — Wounds and Injuries; Neoplastic Processes

STUDY DESIGN:
Intervention Model Description: All subjects will undergoing posterior thoracolumbar arthrodesis procedures utilizing pedicle screw instrumentation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1 (Other): Single Arm. All participants undergoing posterior thoracolumbar arthrodesis procedures betweenT2-S1 in which preplanning is done using the Mazor X robotic system.
  Interventions: Device: Pedicle screw instrumentation using Mazor X robotic system

INTERVENTIONS:
Device: Pedicle screw instrumentation using Mazor X robotic system — Pedicle screw instrumentation using Mazor X robotic system

SUMMARY:
The purpose of the study is to assess screw deviation from pre-planned trajectory using the Mazor X robotic system in patients undergoing posterior thoracolumbar arthrodesis procedures between T2-S1.

DETAILED DESCRIPTION:
This trial will prospectively evaluate screw deviation from pre-planned trajectory using the standard of care Mazor X robotic system. Patients undergoing posterior thoracolumbar arthrodesis procedures utilizing pedicle screw instrumentation at previously uninstrumented levels for degenerative conditions, spinal deformity, spinal infection, trauma, or neoplastic processes between T2-S1 will be asked to participate in this prospective cohort study.

This single centered study will enroll up to 50 patients to achieve a total number of 250 screws for assessment. Subjects will be followed till discharge following surgery. All subjects enrolled in the study will be recruited from a pool of subjects eligible for posterior thoracolumbar arthrodesis surgery.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Degenerative conditions, spinal deformity, spinal infection, traumatic injuries, or neoplastic processes between T2-S1 necessitating placement of pedicle screw instrumentation.
* Surgery performed at The Ohio State University Wexner Medical Center (OSUWMC) via one of the study investigators

Exclusion Criteria:

* Current or previous spinal tumor
* Severe co-morbidities (e.g., heart, respiratory, or renal disease)
* Concurrent involvement in another investigational drug or device study that could confound study data
* Subjects who are pregnant
* Prisoner
* Subjects who do not speak English Relative Exclusion Criteria
* Prior pedicle screw instrumentation at that level (i.e. prior L4-5 instrumentation, now undergoing an L4-S1 fusion, only new S1 screw accuracy would be evaluated in this patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Total deviation (mm) from the pre-planned screw entry point | study completion average 2years
  Total deviation (mm) from the pre-planned screw entry point includes: deviation in angle of insertion in the axial plane (degrees), and deviation in angle of insertion in the sagittal plane (degrees) from an O-arm spin after screw placement.

SECONDARY OUTCOMES:
Accuracy assessment for degree of pedicle breach | 6 weeks post surgery
  The secondary outcome will include traditional accuracy assessment for degree of pedicle breach utilizing the Gertzbein and Robbins classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center Neurological Surgery, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carl AL, Tromanhauser SG, Roger DJ. Pedicle screw instrumentation for thoracolumbar burst fractures and fracture-dislocations. Spine (Phila Pa 1976). 1992 Aug;17(8 Suppl):S317-24. doi: 10.1097/00007632-199208001-00018. PMID 1523519
- [Background] Rose PS, Lenke LG, Bridwell KH, Mulconrey DS, Cronen GA, Buchowski JM, Schwend RM, Sides BA. Pedicle screw instrumentation for adult idiopathic scoliosis: an improvement over hook/hybrid fixation. Spine (Phila Pa 1976). 2009 Apr 15;34(8):852-7; discussion 858. doi: 10.1097/BRS.0b013e31818e5962. PMID 19365256
- [Background] Hyun SJ, Kim KJ, Jahng TA, Kim HJ. Minimally Invasive Robotic Versus Open Fluoroscopic-guided Spinal Instrumented Fusions: A Randomized Controlled Trial. Spine (Phila Pa 1976). 2017 Mar 15;42(6):353-358. doi: 10.1097/BRS.0000000000001778. PMID 27398897
- [Background] Jiang B, Pennington Z, Zhu A, Matsoukas S, Ahmed AK, Ehresman J, Mahapatra S, Cottrill E, Sheppell H, Manbachi A, Crawford N, Theodore N. Three-dimensional assessment of robot-assisted pedicle screw placement accuracy and instrumentation reliability based on a preplanned trajectory. J Neurosurg Spine. 2020 May 29;33(4):519-528. doi: 10.3171/2020.3.SPINE20208. Print 2020 Oct 1. PMID 32470927
- [Background] Gertzbein SD, Robbins SE. Accuracy of pedicular screw placement in vivo. Spine (Phila Pa 1976). 1990 Jan;15(1):11-4. doi: 10.1097/00007632-199001000-00004. PMID 2326693
- [Background] Heary RF, Bono CM, Black M. Thoracic pedicle screws: postoperative computerized tomography scanning assessment. J Neurosurg. 2004 Apr;100(4 Suppl Spine):325-31. doi: 10.3171/spi.2004.100.4.0325. PMID 15070139
- [Background] Wiesner L, Kothe R, Ruther W. Anatomic evaluation of two different techniques for the percutaneous insertion of pedicle screws in the lumbar spine. Spine (Phila Pa 1976). 1999 Aug 1;24(15):1599-603. doi: 10.1097/00007632-199908010-00015. PMID 10457581
- [Background] Rampersaud YR, Pik JH, Salonen D, Farooq S. Clinical accuracy of fluoroscopic computer-assisted pedicle screw fixation: a CT analysis. Spine (Phila Pa 1976). 2005 Apr 1;30(7):E183-90. doi: 10.1097/01.brs.0000157490.65706.38. PMID 15803068
- [Background] van Dijk JD, van den Ende RP, Stramigioli S, Kochling M, Hoss N. Clinical pedicle screw accuracy and deviation from planning in robot-guided spine surgery: robot-guided pedicle screw accuracy. Spine (Phila Pa 1976). 2015 Sep 1;40(17):E986-91. doi: 10.1097/BRS.0000000000000960. PMID 25943084